CLINICAL TRIAL: NCT05178316
Title: A Multicenter Phase 2, 12-week Double-blind, Placebo-controlled, Randomized, Parallel-group Study of JZP150 for the Treatment of Posttraumatic Stress Disorder
Brief Title: A Study of JZP150 in Adults With Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JZP150-201
Record Dates: First submitted 2021-12-08; First posted 2022-01-05 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder; JZP150
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- JZP150 0.3 mg (Experimental): Participants who will be randomized to receive JZP150 0.3 mg orally once daily for up to 12 weeks.
  Interventions: Drug: JZP150
- JZP150 4.0 mg (Experimental): Participants who will be randomized to receive JZP150 4.0 mg orally once daily for up to 12 weeks.
  Interventions: Drug: JZP150
- Placebo (Placebo Comparator): Participants who will be randomized to receive placebo orally once daily for up to 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JZP150 — Oral administration of JZP150 once daily in the morning
  Arms: JZP150 0.3 mg; JZP150 4.0 mg
Drug: Placebo — Oral administration of placebo once daily in the morning
  Arms: Placebo

SUMMARY:
This is a 12-week, double-blind, placebo-controlled, randomized, parallel-group, multicenter study of the safety and efficacy of JZP150 in the treatment of adult participants with post-traumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
JZP150 is an oral, highly selective inhibitor of fatty acid amide hydrolase (FAAH). In this phase 2 study, participants with PTSD will receive either placebo or 1 of 2 doses of JZP150. The primary objective of the study will assess the change in PTSD symptoms from baseline to Week 12 using the Clinician Administered PTSD Scale (CAPS-5).

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 70 years
* Participants must be outpatients with a primary diagnosis of Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) defined PTSD confirmed by the clinical interview
* PTSD is primary diagnosis

Exclusion Criteria:

* Acute or unstable medical condition, behavioral or psychiatric disorder (other than PTSD)
* Suicidal behavior in the past 2 years or active suicidal ideation in the past 6 months
* Ongoing traumatic event or exposure to a traumatic event <3 months prior to Screening
* Index event > 12 years
* Index event is combat trauma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (52):
  - NoesisPharma LLC, Phoenix, Arizona
  - Sanro Clinical Research Group, LLC, Bryant, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Clinical Innovations Inc., Bellflower, California
  - Southern California Research, LLC, Beverly Hills, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Excell Research, Oceanside, California
  - NRC Research Institute, Orange, California
  - CITrials, Riverside, California
  - Clinical Innovations Inc., Santa Ana, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Pacific Clinical Research Management Group LLC, Upland, California
  - MCB Clinical Research Center, Colorado Springs, Colorado
  - CT Clinical Research, Cromwell, Connecticut
  - Yale Center for Clinical Investigation: Church Street Research Unit (CSRU), New Haven, Connecticut
  - Howard University Hospital, Clinical Research Unit, Washington D.C., District of Columbia
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Accel Research Sites -Lakeland Clinical Research Unit, Lakeland, Florida
  - Accel Research Sites Network-St. Petersburg Clinical Research Unit, Largo, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - EZY Medical Research Co, Miami, Florida
  - Behavioral Clinical Research, Inc, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Advanced Discovery Research, Atlanta, Georgia
  - CenExel iResearch, Decatur, Georgia
  - American Medical Research, Inc, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Clinical Trial, Boston, Massachusetts
  - Alivation Research, LLC, Lincoln, Nebraska
  - Altea Research Institute, Las Vegas, Nevada
  - Global Medical Institutes, LLC: Princeton Medical Institute, Princeton, New Jersey
  - SPRI Clinical Trials, Brooklyn, New York
  - Manhattan Behavioral Medicine, Manhattan, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Neuro-Behavioral Clinical Research, Inc, North Canton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Suburban Research Associates, West Chester, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Dell Medical School Universityof Texas at Austin, Austin, Texas
  - Austin Clinical Trial Partners, Austin, Texas
  - Houston Clinical Trials, Bellaire, Texas
  - Relaro Medical Trials, LLC, Dallas, Texas
  - Northpointe Psychiatry, Flower Mound, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Eastside Therapeutic Resource, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 282 participants who met all inclusion criteria and no exclusion criteria were randomized to treatment. Of those 282 participants, 277 received at least 1 dose of study intervention. Five participants did not receive any treatment.
Groups:
- JZP150 0.3 mg: Participants who were randomized to JZP150 0.3 mg orally once daily for up to 12 weeks.
- JZP150 4.0 mg: Participants who were randomized to JZP150 4.0 mg orally once daily for up to 12 weeks.
- Placebo: Participants who were randomized to placebo orally once daily for up to 12 weeks.
Period: Overall Study
Arm/Group | JZP150 0.3 mg | JZP150 4.0 mg | Placebo
Started | 55 | 113 | 109
Completed | 38 | 74 | 78
Not Completed | 17 | 39 | 31
Not completed — Adverse Event | 5 | 4 | 9
Not completed — Enrolled in Error | 1 | 2 | 1
Not completed — Lost to Follow-up | 3 | 15 | 11
Not completed — Noncompliance | 1 | 3 | 1
Not completed — Other | 0 | 1 | 0
Not completed — Physician Decision | 0 | 3 | 2
Not completed — Protocol deviation | 1 | 0 | 1
Not completed — Sponsor decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 11 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | JZP150 0.3 mg | JZP150 4.0 mg | Placebo | Total
Number analyzed (Participants) | 54 | 113 | 110 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (13.54) | 38.6 (12.45) | 41.2 (12.52) | 39.6 (12.72)
Age, Customized [Count of Participants; unit: Participants] — Population: Age Group 1 was assessed in the Safety Analysis Set.
  Participants
    ≤65 years | 53 | 111 | 106 | 270
    >65 years | 1 | 2 | 4 | 7
Age, Customized [Count of Participants; unit: Participants] — Population: Age Group 2 was assessed in the Safety Analysis Set.
  Participants
    ≤45 years | 37 | 79 | 72 | 188
    >45 years | 17 | 34 | 38 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 85 | 81 | 210
  Male | 10 | 28 | 29 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 3 | 6 | 12
  Black or African American | 12 | 16 | 15 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  White | 38 | 92 | 85 | 215
  Declined to state | 1 | 2 | 0 | 3
  Multiple | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 12 in Clinician Administered Posttraumatic Stress Disorder (PTSD) Scale (CAPS-5) Total Symptom Severity Score
Description: Clinician Administered Posttraumatic Stress Disorder (PTSD) Scale (CAPS-5) is a clinician administered, clinical interview where participants report on their symptoms of PTSD on a scale. The CAPS-5 total score ranges between 0 and 80. Higher scores indicate more severe PTSD symptoms.
  Change in CAPS-5 total score is being reported, where negative mean scores indicate an improvement in clinical outcome.
Time Frame: Baseline to Week 12
Population: CAPS-5 total symptom severity score was assessed in participants with available data in the Full Analysis Set 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JZP150 0.3 mg | JZP150 4.0 mg | Placebo
Number analyzed (Participants) | 44 | 79 | 85
score on a scale | -17.0 (13.75) | -17.8 (12.59) | -17.6 (11.99)
Statistical Analysis 1: Comparison: JZP150 0.3 mg vs Placebo; Test type: Superiority; p = 0.8862, Mixed Models Analysis; Least squares mean difference = 0.31, 95% CI 2-sided [-3.98 to 4.60], Standard Error of Mean 2.175
Statistical Analysis 2: Comparison: JZP150 4.0 mg vs Placebo; Test type: Superiority; p = 0.6832, Mixed Models Analysis; Least squares mean difference = -0.74, 95% CI 2-sided [-4.32 to 2.84], Standard Error of Mean 1.817

2. Secondary Outcome: Mean Change From Baseline to Week 12 in Clinical Global Impression of Severity (CGI-S)
Description: Clinical Global Impression of Severity (CGI-S) is a clinician assessment used to assess the severity of the participants' PTSD on a scale range of 1 to 7, where 1 indicates "normal, not at all ill" and a 7 indicates "among the most extremely ill participants".
  Change in CGI-S is being reported with negative mean values indicating an improvement in clinical outcome.
Time Frame: Baseline to Week 12
Population: CGI-S was assessed in participants with available data in the Full Analysis Set 1 (defined as
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JZP150 0.3 mg | JZP150 4.0 mg | Placebo
Number analyzed (Participants) | 44 | 82 | 85
score on a scale | -1.4 (1.10) | -1.3 (1.27) | -1.2 (1.08)
Statistical Analysis 1: Comparison: JZP150 0.3 mg vs Placebo; Test type: Superiority; p = 0.4522, Mixed Models Analysis; Least squares mean difference = -0.15, 95% CI 2-sided [-0.55 to 0.25], Standard Error of Mean 0.204
Statistical Analysis 2: Comparison: JZP150 4.0 mg vs Placebo; Test type: Superiority; p = 0.2032, Mixed Models Analysis; Least squares mean difference = -0.22, 95% CI 2-sided [-0.55 to 0.12], Standard Error of Mean 0.169

3. Secondary Outcome: Mean Change From Baseline to Week 12 in Patient Global Impression of Severity (PGI-S)
Description: Patient Global Impression of Severity (PGI-S) is a patient assessment designed to evaluate severity of PTSD symptoms on a scale from 1 to 5, where 1 indicates "none" and 5 indicates "very severe".
  Change in PGI-S is being reported with negative mean values indicating an improvement in clinical outcome.
Time Frame: Baseline to Week 12
Population: PGI-S was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JZP150 0.3 mg | JZP150 4.0 mg | Placebo
Number analyzed (Participants) | 44 | 81 | 85
score on a scale | -1.0 (1.17) | -1.1 (1.11) | -1.0 (1.09)
Statistical Analysis 1: Comparison: JZP150 0.3 mg vs Placebo; Test type: Superiority; p = 0.7170, Mixed Models Analysis; Least squares mean difference = -0.06, 95% CI 2-sided [-0.38 to 0.26], Standard Error of Mean 0.165
Statistical Analysis 2: Comparison: JZP150 4.0 mg vs Placebo; Test type: Superiority; p = 0.2423, Mixed Models Analysis; Least squares mean difference = -0.16, 95% CI 2-sided [-0.43 to 0.11], Standard Error of Mean 0.137

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to Week 12.
Description: Due to the receipt of the incorrect intervention, 1 participant who was randomized to the JZP150 0.3 mg arm actually received placebo as their first dose, and thus was analyzed in the JZP150 0.3 mg arm for the Full Analysis Set 2 and in the placebo arm for the Safety Analysis Set.
Arm/Group | JZP150 0.3 mg | JZP150 4.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/113 | 0/110
Serious Adverse Events (participants affected / at risk) | 1/54 | 2/113 | 1/110
Other Adverse Events (participants affected / at risk) | 20/54 | 30/113 | 24/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JZP150 0.3 mg (N=54) | JZP150 4.0 mg (N=113) | Placebo (N=110)
Seizure (Nervous system disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JZP150 0.3 mg (N=54) | JZP150 4.0 mg (N=113) | Placebo (N=110)
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 10
Nausea (Gastrointestinal disorders) | 3 | 8 | 4
Fatigue (General disorders) | 3 | 4 | 3
Dizziness (Nervous system disorders) | 3 | 4 | 0
Headache (Nervous system disorders) | 4 | 8 | 6
Somnolence (Nervous system disorders) | 3 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT05178316/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT05178316/SAP_001.pdf